CLINICAL TRIAL: NCT00145678
Title: Psychodynamic Therapy for Patients With Borderline Personality Disorder and Alcohol Abuse
Brief Title: Psychodynamic Therapy For Co-occurring Borderline Personality Disorder and Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUNY UMU IRB 4968; 130230-44
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Borderline Personality Disorder; Alcohol Use Disorder
Keywords: borderline; alcohol; substance; psychodynamic; psychotherapy; psychoanalytic
MeSH Terms: conditions — Borderline Personality Disorder; Alcoholism | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dynamic deconstructive psychotherapy (Experimental): weekly individual psychotherapy of 50 minute duration lasting 12-18 months
  Interventions: Behavioral: Psychodynamic Therapy
- optimized community care (Active Comparator): eclectic weekly individual and group psychotherapy, as well as drug and alcohol rehabilitation
  Interventions: Behavioral: Optimized Community Care

INTERVENTIONS:
Behavioral: Psychodynamic Therapy — Dynamic deconstructive psychotherapy is a time-limited (12-18 month) manual-based form of psychodynamic therapy that aims to remediate specific neurocognitive capacities responsible for processing of emotional experiences.
  Other Names: Dynamic Deconstructive Psychotherapy
  Arms: dynamic deconstructive psychotherapy
Behavioral: Optimized Community Care — individual and group psychotherapy in a private practice, clinic, and/or rehab setting, with an eclectic orientation
  Other Names: Treatment as Usual
  Arms: optimized community care

SUMMARY:
The purpose of the study is to determine the feasibility and effectiveness of a modified form of psychodynamic psychotherapy for persons suffering from co-occurring borderline personality disorder and an alcohol use disorder.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a condition that can cause significant distress and increased risk of death. Many persons with BPD also have an alcohol use disorder (AUD) and there is evidence that this can worsen the outcome and course of both disorders.

A manual-based form of psychodynamic therapy (PT), labeled dynamic deconstructive psychotherapy, has been developed for particularly challenging patients with BPD, especially those with co-occurring substance use disorders. It aims to remediate specific neurocognitive capacities that are responsible for processing of emotional experiences, and so diminishes symptoms of BPD and promotes the development of a coherent and differentiated self-structure. PT has been shown to be helpful for BPD, but has not been tested for people who have BPD with co-occurring substance use disorders.

The proposed study is a randomized controlled trial of PT for persons with BPD and co-occurring AUD that will generate some initial data that can be used to determine the need and feasibility for further outcome studies. Participants are randomized to either a study group receiving weekly PT or to a control group receiving usual care. Enrollment is 15 participants in each group. The study group will receive 12-18 months of PT, with naturalistic follow-up. Outcome measures are administered by a research assistant at enrollment, 3 months, 6 months, 9 months, 12 months, and 30 months.

The investigators anticipate that the PT group will show trends towards better retention in treatment and greater reduction in parasuicides, alcohol misuse, and institutional care. If so, this would have important and positive implications for the large group of patients who suffer from BPD and co-occurring AUD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Meets diagnostic criteria for borderline personality disorder and for active alcohol abuse or dependence
* At least average intelligence

Exclusion Criteria:

* Meets diagnostic criteria for schizophrenia, or schizoaffective disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
episodes of parasuicide, alcohol intoxication, institutional care | 12 months

SECONDARY OUTCOMES:
depression, dissociation, core symptoms of borderline pd, perceived social support | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Gregory, M.D., Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, University Hospital, Syracuse, New York, United States

REFERENCES:
- [Background] Gregory RJ. Thematic stages of recovery in the treatment of borderline personality disorder. Am J Psychother. 2004;58(3):335-48. doi: 10.1176/appi.psychotherapy.2004.58.3.335. PMID 15675256
- [Background] Gregory RJ. Borderline attributions. Am J Psychother. 2007;61(2):131-47. doi: 10.1176/appi.psychotherapy.2007.61.2.131. PMID 17760318
- [Background] Gregory RJ. The deconstructive experience. Am J Psychother. 2005;59(4):295-305. doi: 10.1176/appi.psychotherapy.2005.59.4.295. PMID 16555459
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793